CLINICAL TRIAL: NCT06700993
Title: Suicide Treatment and Recovery in Integrated Behavioral Health (STRIBH)
Acronym: STRIBH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate Comtois, Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00016520; P50MH129708 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Suicidal Ideation and Behavior
MeSH Terms: conditions — Suicidal Ideation; Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Partnering primary care clinics will recruit study participants and provide them treatment as usual in their Collaborative Care or other Integrated Behavioral Health program. This will be followed by training in the experimental intervention, the Connections model. Trained clinicians will recruit study participants and provide them with the Connections model in their Collaborative Care or other Integrated Behavioral Health program. This is a pilot study in preparation for a larger stepped wedge or other cluster randomized trial.
Who Masked: Outcomes Assessor
Masking Description: All outcomes are completed through surveys so the research team is not blinded, per se, but they are not involved in the participant responses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (Experimental)
  Interventions: Behavioral: Connections model
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual in Collaborative Care or Integrated Behavioral Health

INTERVENTIONS:
Behavioral: Treatment as Usual in Collaborative Care or Integrated Behavioral Health — Treatment as Usual will be whatever primary care and behavioral health services are standardly implemented for adolescents or young adults experiencing suicidality
  Arms: Treatment as Usual
Behavioral: Connections model — The Connections model applies the Aeschi Model of suicide care to Collaborative Care or other Integrated Behavioral Health by centering the patient's clinical narrative, focusing treatment on the patient's unique drivers of suicide, and maximizing collaboration while maintaining the standards of suicide assessment and management expected by accrediting bodies.
  Arms: Experimental Condition

SUMMARY:
The suicide rate has increased 28% over the past two decades while heart disease, diabetes, and cancer mortality has declined. Starting in 2011, new standards have led to improved adoption and reach of suicide risk surveillance in primary and specialty care. Treatment, however, has lagged. Collaborative Care in primary care settings has demonstrated small but significant reductions in suicidal ideation when a recognized psychological treatment model is included but not when Collaborative Care only includes medication management, suggesting that improvements to psychological treatments in Collaborative Care could further improve suicide outcomes. Developed in a series of conferences in Aeschi Switzerland, the "Aeschi Model" based on the clinical narrative has become an established approach to suicide care endorsed by leaders across the suicidology field - including the developers of major evidence-based suicide interventions. With support from the Methods Core, this Exploratory (R34) study of the University of Washington Suicide Care Research Center (SCRC) will co-design and pilot test the "Connections model" that integrates Aeschi Model with Collaborative Care or other Integrated Behavioral Health with adolescent and young adult patients (age 13-30 years) who do not require immediate crisis intervention. This study will focus on increasing therapeutic alliance - a key proposed mechanism of the Aeschi approach and the SCRC. The aims of this study are to partner with diverse primary care clinics to conduct a pilot test of the Connections model compared to treatment as usual in six primary care clinics to determine (a) usability and acceptability of the intervention components to patients and providers and (b) the components' potential impact on therapeutic alliance and patient and provider self-efficacy, and (c) potential impact on suicidal outcomes. Given the strong theoretical basis for both the Aeschi Model and Collaborative Care, this proposal has the potential to develop a high impact intervention that will both reduce suicide risk and improve therapeutic alliance - potentially without any increase in the quantity of care.

DETAILED DESCRIPTION:
This study will focus on increasing therapeutic alliance - a key proposed mechanism of the Aeschi approach and the SCRC. The aims of this study are to partner with diverse primary care clinics to conduct a pilot test of the Connections model compared to treatment as usual in six primary care clinics to determine (a) usability and acceptability of the intervention components to patients and providers and (b) the components' potential impact on therapeutic alliance and patient and provider self-efficacy, and (c) potential impact on suicidal outcomes. Given the strong theoretical basis for both the Aeschi Model and Collaborative Care, this proposal has the potential to develop a high impact intervention that will both reduce suicide risk and improve therapeutic alliance - potentially without any increase in the quantity of care.

ELIGIBILITY:
Inclusion Criteria:

* 13-30 years of age, experiencing suicidal thoughts or attempted suicide in the past year, not requiring immediate crisis care (as determined by the UW Primary Care team), not enrolled in specialty behavioral health treatment, can read one of the 4 most common languages in Seattle (English, Spanish, Chinese, or Vietnamese), enrolled in a primary care clinic with an integrated behavioral health provider available to see them, and ability to consent to participate.

Exclusion Criteria:

* any clinical medical/psychiatric condition, severity of that condition, or life situation that, in the opinion of the primary care or research team, compromises safe and voluntary study participation (e.g., high risk for suicide requiring transfer to higher level of care; physically aggressive, custody conflict)

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | baseline, one month, and two months
  Four item scale to measure the acceptability of an intervention
System Usability Scale | baseline, one month, and two months
  The System Usability Scale is a 10-item measure of the usability of a tool, and is considered the industry standard for measuring usability in the UCD field. A SUS score of 80 is generally seen as a threshold for a highly usable system.
Harkavy-Asnis Suicide Scale | baseline, one month and two months
  This measure assesses the frequency of suicidal ideation on a 5-point Likert scale, with 0 indicating "never" and 4 indicating "most or all of the time". Higher scores reflect higher severity and frequency of suicidal ideation.

OTHER OUTCOMES:
The Columbia Suicide Severity Rating Scale Screener (C-SSRS) | baseline, one month and two months
  A measure of suicidal thoughts and behaviors. Suicide ideation is rated on a scale of 1 to 5, with higher numbers reflecting more severe ideation. Suicidal behaviors are count measures, with higher numbers reflecting more attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Comtois, PhD, MPH, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: Undecided